CLINICAL TRIAL: NCT02606097
Title: A Phase 2 Study of Regorafenib in Metastatic Gastrointestinal Stromal Tumours With C-KIT exon17 Mutation
Brief Title: Regorafenib in GIST With Secondary C-KIT Exon 17 Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yeh Chun-Nan, Professor and Chief, Department of Surgery, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17298
Record Dates: First submitted 2015-11-12; First posted 2015-11-17 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Gastrointestinal Stromal Tumour (GIST)
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- regorafenib (Experimental): regorafenib 160 mg daily, 3 weeks on/1 week off
  Interventions: Drug: regorafenib

INTERVENTIONS:
Drug: regorafenib
  Other Names: stivarga

SUMMARY:
The main purpose of this study is to examine whether regorafenib treatment can help people with gastrointestinal stromal tumours (GIST) and have gene mutation on c-kit exon 17. The safety of regorafenib treatment is also examined.

ELIGIBILITY:
Inclusion Criteria:

An eligible subject must fulfill all of the following inclusion criteria:

* Signed informed consent (IC) obtained before any study specific procedure. Patients must be able to understand and willing to sign the written IC.
* Pathologically confirmed gastrointestinal stromal tumours.
* All patients had received imatinib or sunitinib.
* Pathological confirmed c-kit exon 17 mutation.
* At least one measurable lesion in a non-irradiated area or allowed to be tracked whether there are circumstances recurrence by computed tomography (CT) or magnetic resonance imaging (MRI).
* Aged > 20 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Life expectancy greater than 12 weeks.
* Adequate bone marrow function: 1) Absolutely neutrophil count >= 1.5 x10^9/L or white blood cell count (WBC) >= 4x10^9/L; 2) Hemoglobin >= 9 g/dL; 3) Platelet count >= 100x10^9/L.
* Adequate liver function: 1) Total bilirubin <= 1.5x the upper limit of normal (ULN); 2) Alanine Aminotransferase (ALT) & Aspartate Aminotransferase (AST) <= 2.5x ULN if without liver metastasis or <= 5x ULN if with hepatic metastasis; 3) Alkaline phosphatase <= 2.5x ULN if without liver metastasis or <= 5x ULN if with hepatic metastasis or bone metastasis; 4) Bilirubin < 2x ULN.
* Adequate renal function: creatinine <1.5x ULN.
* Patients must be accessible for treatment and follow-up in the participating centers.

Exclusion Criteria:

Subject will not meet any of the following exclusion criteria:

* Major surgery within four weeks prior to entering the study.
* Patients with central nervous system (CNS) metastasis, including clinical suspicion.
* Patients who are under active or uncontrolled infections.
* Patients who with unstable angina (angina symptoms at rest, new-onset angina (begun within the last 3 months) or myocardial infarction history 6 months before entry.
* Cardiac arrhythmia requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
* Congestive heart failure New York Heart Association (NYHA) class 2.
* Uncontrolled hypertension (systolic blood pressure [BP] > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management.
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before the start of study medication.
* Patients who are pregnant or with breast feeding.
* Other concomitant or previously malignancy within 5 years except for in situ cervix cancer or squamous cell carcinoma of the skin treated by surgery only.
* Mental status is not fit for clinical trial.
* Cannot take study medication orally.
* Fertile men and women unless using a reliable and appropriate contraceptive method.
* Patients with evidence or history of any bleeding diathesis, irrespective of severity.
* Any hemorrhage or bleeding event >= Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 within 4 weeks prior to the start of study medication.
* Non-healing wound, ulcer, or bone fracture.
* Renal failure requiring hemo-or peritoneal dialysis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Overall clinical benefit rate | till 2 weeks after last dose
  complete response (CR), partial response (PR), and stable disease (SD)

SECONDARY OUTCOMES:
Progression free survival (PFS) | till study end, estimated 3 years
Overall survival (OS) | till study end, estimated 3 years

OTHER OUTCOMES:
Adverse events (AEs) | till 2 weeks after last dose
  Incidence of AEs will be shown and severity will be graded using NCI-CTCAE version 4.0
Changes in clinical hematology laboratory result by hemoglobin (Hb) | till 2 weeks after last dose
  (unit: g/dL)
Changes in clinical hematology laboratory result by hematocrit (Hct) | till 2 weeks after last dose
  (unit: %)
Changes in clinical hematology laboratory result by platelet count | till 2 weeks after last dose
  (unit: 10^9/L)
Changes in clinical hematology laboratory result by red blood cell (RBC) count | till 2 weeks after last dose
  (unit: 10^9/L)
Changes in clinical hematology laboratory result by white blood cell (WBC) count | till 2 weeks after last dose
  (unit: 10^9/L)
Clinical hematology laboratory result by WBC differential | till 2 weeks after last dose
  (unit: %)
Changes in clinical biochemistry laboratory result by potassium level | till 2 weeks after last dose
  (unit: mmol/L)
Changes in clinical biochemistry laboratory result by calcium level | till 2 weeks after last dose
  (unit: mmol/L)
Changes in clinical biochemistry laboratory result by glucose level | till 2 weeks after last dose
  (unit: mmol/L)
Changes in clinical biochemistry laboratory result by lactate dehydrogenase (LDH) level | till 2 weeks after last dose
  (unit: U/L)
Changes in clinical biochemistry laboratory result by blood urea nitrogen (BUN) level | till 2 weeks after last dose
  (unit: mmol/L)
Changes in clinical biochemistry laboratory result by creatinine level | till 2 weeks after last dose
  (unit: mg/dL)
Changes in clinical biochemistry laboratory result by total and direct bilirubin levels | till 2 weeks after last dose
  (unit: mg/dL)
Changes in clinical biochemistry laboratory result by albumin levels | till 2 weeks after last dose
  (unit: g/L)
Changes in clinical biochemistry laboratory result by alanine aminotransferase(ALT) levels | till 2 weeks after last dose
  (unit: U/L)
Changes in clinical biochemistry laboratory result by aspartate aminotransferase (AST) levels | till 2 weeks after last dose
  (unit: U/L)
Changes in clinical biochemistry laboratory result by alkaline phosphatase (ALP) level | till 2 weeks after last dose
  (unit: U/L)
Changes in clinical biochemistry laboratory result by thyroid-stimulating hormone (TSH) level | till 2 weeks after last dose
  (unit: mIU/L)
Changes in clinical biochemistry laboratory result by T3 level | till 2 weeks after last dose
  (unit: mIU/L)
Changes in clinical biochemistry laboratory result by T4 level | till 2 weeks after last dose
  (unit: mIU/L)
Changes in clinical urinalysis result by WBC count | till 2 weeks after last dose
  (unit: 10^9/L)
Changes in clinical urinalysis result by RBC count | till 2 weeks after last dose
  (unit: 10^9/L)
Changes in clinical urinalysis result by pH level | till 2 weeks after last dose
Changes in clinical urinalysis result by protein level | till 2 weeks after last dose
Changes in clinical urinalysis result by glucose level | till 2 weeks after last dose
  (unit: mmol/L)
Changes in clinical coagulation results by prothrombin time (PT) | till 2 weeks after last dose
  (unit: sec)
Changes in clinical coagulation results by activated partial thromboplastin time (APTT) | till 2 weeks after last dose
  (unit: sec)
Changes in clinical coagulation results by international normalized ratio (INR) | till 2 weeks after last dose
Physical examination | till 2 weeks after last dose
Changes in vital signs by respiratory rate | till 2 weeks after last dose
  (unit: times/min)
Changes in vital signs by pulse rate | till 2 weeks after last dose
  (unit: times/min)
Changes in vital signs by systolic blood pressure | till 2 weeks after last dose
  (unit: mmHg)
Changes in vital signs by diastolic blood pressure | till 2 weeks after last dose
  (unit: mmHg)
Changes in vital signs by body temperature | till 2 weeks after last dose
  (unit: degree celsius)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Nan Yeh, MD, Principal Investigator — Professor and Chief, Department of Surgery
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Yeh CN, Chen MH, Chen YY, Yang CY, Yen CC, Tzen CY, Chen LT, Chen JS. A phase II trial of regorafenib in patients with metastatic and/or a unresectable gastrointestinal stromal tumor harboring secondary mutations of exon 17. Oncotarget. 2017 Jul 4;8(27):44121-44130. doi: 10.18632/oncotarget.17310. PMID 28487491